CLINICAL TRIAL: NCT02829086
Title: Evaluation of the U.S. Committee for Refugees and Immigrants (USCRI): Refugee Family Strengthening (RFS) Program
Brief Title: Evaluation of the Refugee Family Strengthening (RFS) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Committee for Refugees and Immigrants (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 90FM0092-01-00
Record Dates: First submitted 2016-06-29; First posted 2016-07-12 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Financial Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group I (Experimental): Participants in Group I will receive the following interventions: Intro to Relationship Enhancement (8 hours), Family Stress and Conflict Management (8 hours), and case management
  Interventions: Other: Relationship Enhancement; Other: Family Stress and Conflict Management
- Group II (Experimental): Participants in Group II will receive the following interventions: Intro to Relationship Enhancement (8 hours), RE & Financial Management (8 hours), and case management
  Interventions: Other: Relationship Enhancement; Other: Financial Management
- Group III (No Intervention): Participants in Group III will receive the the standard care of all participants, case management ONLY

INTERVENTIONS:
Other: Relationship Enhancement — Relationship Enhancement is a curriculum based program provided by a facilitator over an 8 hour skill-based education intervention.
  Arms: Group I; Group II
Other: Family Stress and Conflict Management — Family Stress and Conflict Management is a curriculum based program provided by a facilitator over an 8 hour skill-based education intervention.
  Arms: Group I
Other: Financial Management — Family Management is a curriculum based program provided by a facilitator over an 8 hour skill-based education intervention.
  Arms: Group II

SUMMARY:
The US Committee for Refugees and Immigrants (USCRI) will be conducting an evaluation of a healthy marriage and relationship program developed by USCRI titled Refugee Family Strengthening (RFS) Program. This program is funded through an initiative of the Administration for Children and Families, Office of Family Assistance (OFA).

The study is intended to measure if the identified interventions improve the well-being of individuals and families within the refugee and immigrant population served by USCRI. Outcomes to be measured include behavioral outcomes and perceptual changes towards healthy relationships, family development, and positive home environment. The study will examine the following:

1. Participants will identify utilizing healthy marriage and relationship skills.
2. Participants will report an increase in satisfaction with conflict management with others after completion of the relationship workshop series.
3. Participants will report an increase in quality and time spent with children.
4. Participants will report an increase in economic stability.

DETAILED DESCRIPTION:
The US Committee for Refugees and Immigrants (USCRI) will be conducting an evaluation of a healthy marriage and relationship program developed by USCRI titled Refugee Family Strengthening (RFS) Program. This program is funded through an initiative of the Administration for Children and Families, Office of Family Assistance (OFA).

The Refugee Family Strengthening (RFS) Program builds on literature and existing research from the healthy marriage and relationship initiatives developed by ACF over the last 10 years, in particular the Supporting Healthy Marriage Program initiative that established a randomized clinical trial. In addition, marriage and relationship education/ enrichment literature and research has expanded dramatically over the past 35 years. The most glaring shortcoming of this database is the limited types of populations that are sampled and included in studies. USCRI's RFS program will provide important data about a diverse group of subjects that is currently unavailable.

The aim of the evaluation is to determine the effect of participating in two interventions on the population of refugee and immigrant couples, families, and individuals, served by USCRI. The program will target individuals ages 16 and older using a randomized control design. The program will be implemented with individuals, couples, and families. RFSP will recruit 9,350 individuals over the 5 year tenure of the project, 3115 of which will serve as control subjects, the remaining 6,235 subjects will be randomly assigned to intervention groups at each of the 11 selected sites that are participating in the project. Control subjects will not receive the intervention workshops, only case management.

The intervention is to be delivered as follows:

Group I: Intro to Relationship Enhancement (RE) (8 hours), Family Stress & Conflict Management (8 hours), and case management Group II: Intro to Relationship Enhancement (RE) (8 hours), & Financial Management (8 hours), and case management Group III: Case management ONLY

Data will be collected and analyzed across 3 collection points: Pre-test immediately before the start of the interventions, Post-test immediately upon completion of the interventions, and again at 6 months following the pre-test date.

Results will be analyzed to determine gains towards the following research questions:

When participating in the RFS program:

1. Do individuals who participate in the two RFS interventions demonstrate favorable impact in the four program outcomes as compared to those who participate in the control?
2. What are the differences in gains for subjects who participate in the two different interventions?
3. What are the long-term effects of participation in the RFS interventions on individuals?

The local evaluation is expected to reflect progress toward project outcomes and is anticipated to demonstrate significant results that will be highlighted and prepared for dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Refugee or Immigrant

Exclusion Criteria:

* Individuals under the age of 16
* Individuals that are not identified as refugees or immigrants

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5365 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Healthy Relationship Skills | At program enrollment-during registration, immediately after completing 8 hour Relationship Enhancement intervention and at 6 month follow up.
  Questionnaire developed for intervention to measure change from before 8 hour intervention to after intervention

SECONDARY OUTCOMES:
Conflict Management Skills | At program enrollment-during registration, immediately after completing 8 hour Conflict Resolution intervention and at 6 month follow up.
  Questionnaire developed for intervention to measure change from before 8 hour intervention to after intervention
Economic Stability | At program enrollment-during registration, immediately after completing 8 hour Financial Literacy intervention and at 6 month follow up.
  Questionnaire developed for intervention to measure change from before 8 hour intervention to after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Salerno, DNP, Principal Investigator — Possibilities for Change
Locations (11):
- United States (11):
  - International Institute of Los Angeles, Los Angeles, California
  - USCRI Des Moines, Des Moines, Iowa
  - USCRI Detroit, Dearborn, Michigan
  - Jewish Vocational Services, Kansas City, Missouri
  - International Institute of St. Louis, St Louis, Missouri
  - USCRI Albany, Albany, New York
  - USCRI North Carolina, Raleigh, North Carolina
  - International Institute of Erie, Erie, Pennsylvania
  - Nationalities Services Center, Philadelphia, Pennsylvania
  - YMCA International Services, Houston, Texas
  - Vermont Refugee Resettlement Program, Colchester, Vermont

IPD SHARING:
Plan to Share IPD: Undecided